CLINICAL TRIAL: NCT03951285
Title: Vitamin B3 as a Novel Mitochondrial Therapy for Obesity
Brief Title: Nicotinamide Riboside and Mitochondrial Metabolism
Acronym: VitaPower
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other); University of Iowa (Other); Finnish Institute for Health and Welfare (Other Government); Göteborg University (Other)
Responsible Party: Principal Investigator, Kirsi Pietiläinen, Professor in Clinical Metabolism, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NRtwins_0001
Record Dates: First submitted 2019-01-10; First posted 2019-05-15 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Obesity
Keywords: Obesity; Metabolic syndrome; Vitamin B3; Nicotinamide riboside; Mitochondrial dysfunction; Mitochondria; Adipose tissue; Skeletal muscle
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Mitochondrial Diseases | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: Study with two interventions in healthy monozygotic twin pairs. In the first intervention, both members of BMI-discordant monozygotic twins are treated with Nicotinamide Riboside (NR). With this unique model, the investigators obtain the information on how beneficial NR is in two different BMI classes (obese and leaner) with an identical genomic background. In the second intervention, monozygotic twins concordant for body weight are selected and randomized to treatment. One member of the twin pair is treated with NR while the other co-twin gets placebo. With the twin set-up, the investigators can detect a significant treatment effect, and the heritability of NR treatment can be estimated as well.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NR (Experimental): One intervention includes healthy BMI-discordant monozygotic twin pairs, which both are treated with NR. With this unique model, the investigators obtain the information on how beneficial NR is in two different BMI classes (obese and leaner) with an identical genomic background.
  The final dose for NR will be 1 g/day. The daily NR dose is gradually escalated by 250 mg/week so that the full dose of 1 g/day is reached in one month. The intervention time with the full NR dose is 4 months, total intervention time 5 months. At the end of the study, the daily dose will be decreased by 250 mg/week rate.
  Interventions: Dietary Supplement: NR in BMI-discordant twins; Dietary Supplement: NR in BMI-concordant twins
- Placebo (Placebo Comparator): The second intervention includes monozygotic twins concordant for body weight. It's randomized which member of the twin pair is treated with NR while the other co-twin gets placebo.
  The final dose for placebo will be 1 g/day. The daily placebo dose is gradually escalated by 250 mg/week so that the full dose of 1 g/day is reached in one month. The intervention time with the full placebo dose is 4 months, total intervention time 5 months. At the end of the study, the daily dose will be decreased by 250 mg/week rate.
  Interventions: Dietary Supplement: NR in BMI-concordant twins

INTERVENTIONS:
Dietary Supplement: NR in BMI-discordant twins — Water-soluble form of vitamin B3, nicotinamide riboside (NR) is used in this study. The NR product name is Niagen, produced by ChromaDex. NR does not cause the known side effects (vasodilation and flushing) of another vitamin B3, niacin.
  Other Names: Niagen; Nicotinamide riboside
  Arms: NR
Dietary Supplement: NR in BMI-concordant twins — Water-soluble form of vitamin B3, nicotinamide riboside (NR) is used in this study. The NR product name is Niagen, produced by ChromaDex. NR does not cause the known side effects (vasodilation and flushing) of another vitamin B3, niacin.
  Other Names: Niagen

SUMMARY:
Vitamin B3 has recently been found to be a potent modifier of energy metabolism, especially the function of mitochondria. Mitochondria power up all cells in our bodies, by generating fuel, ATP, for cellular functions. In previous studies, it has been discovered that mitochondrial biogenesis and oxidative metabolism in adipose tissue is severely impaired in obesity, already at a young adult age. Here the investigators describe a proposal where they use nicotinamide riboside (NR), a form of vitamin B3 naturally found in milk, to activate dysfunctional mitochondria, in particular the SIRT/NAD+ pathway, and to rescue signs of obesity-related diseases. The investigators use a unique human study design: monozygotic twins either discordant or concordant for obesity, to examine the effects of NR on mitochondrial function in muscle, adipose tissue and the metabolism of the whole body. The upcoming upcoming results are important for understanding the links between mitochondrial dysfunction and chronic metabolic diseases in humans, as well as for clarifying mechanisms of the novel nutritional therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

1. BMI >18.5 kg/m2 in both members of the twin pair
2. Agreed to maintain current level of physical activity throughout the study
3. Agreed to avoid vitamin supplementation or nutritional products with vitamin B3 14 days prior to the enrolment and during the study
4. Written, informed consent to participate in the study

Exclusion Criteria:

1. Unstable medical conditions as determined by the principal investigator
2. Clinically significant abnormal lab results at screening (e.g. AST and/or ALT > 2 x ULN, and/or bilirubin > 2 x ULN)
3. Subjects who have a planned surgery during the course of the trial
4. History of or a current diagnosis of any cancer (except for successfully treated basal cell carcinoma diagnosed less than 5 years prior to screening). Subjects with cancer in full remission more than 5 years after diagnosis are acceptable.
5. History of blood/bleeding disorders
6. Immunocompromised individuals such as subjects that had undergone organ transplantation or subjects diagnosed with human immunodeficiency virus (HIV)
7. Hepatitis
8. Blood donation in the previous 2 months
9. Anemia (hemoglobin <120)
10. Participation in a clinical research trial within 30 days prior to randomization
11. Allergy or sensitivity to study supplement ingredients
12. Individuals who are cognitively impaired and/or who are unable to give informed consent.
13. Any other condition, which in the principal investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may have posed significant risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Mitochondrial biogenesis - mitochondrial DNA quantification | At baseline and 5 months after supplementation
  Change in amount of mitochondrial DNA in skeletal muscle and adipose tissue (mtDNA quantification)
Mitochondrial biogenesis - mitochondria-related mRNA expression | At baseline and 5 months after supplementation
  Change in mitochondria-related mRNA expression in skeletal muscle and adipose tissue (qPCR)
Mitochondrial biogenesis - electron microscopy | At baseline and 5 months after supplementation
  Change in mitochondria histology by electron microscopy evaluation of skeletal muscle

SECONDARY OUTCOMES:
NAD+ and related metabolite levels in blood | At baseline and 5 months after supplementation
  Change in levels of NAD+ and related metabolites such as: NADP+, nicotinic acid adenine dinucleotide, nicotinamide, and nicotinamide mononucleotide in blood using high performance liquid chromatography-mass spectrometry
Skeletal muscle mitochondrial oxidative capacity | At baseline and 5 months after supplementation
  Change in mitochondrial function in skeletal muscle by immunohistochemical respiratory chain enzyme analysis

OTHER OUTCOMES:
Body weight and body composition | At baseline and 5 months after supplementation
  Change in body weight as well as fat mass and fat free mass measured with bioimpedance and DEXA scanning, fat distribution by magnetic resonance imaging
Ectopic lipid accumulation in liver and muscle (in vivo) | At baseline and 5 months after supplementation
  Change in liver and skeletal muscle lipid accumulation measured with H-MRS in vivo
Whole body insulin sensitivity | At baseline and 5 months after supplementation
  Insulin sensitivity as measured by oral glucose tolerance test (OGTT)-derived indexes
Circulating inflammation markers | At baseline and 5 months after supplementation
  Change in circulating levels of IL-2, IL-5, IL-6, IL-12 and TNF-alpha will be measured by multiplex

CONTACTS AND LOCATIONS:
Overall Officials: Kirsi H Pietiläinen, MD PhD, Principal Investigator — University of Helsinki

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Naukkarinen J, Heinonen S, Hakkarainen A, Lundbom J, Vuolteenaho K, Saarinen L, Hautaniemi S, Rodriguez A, Fruhbeck G, Pajunen P, Hyotylainen T, Oresic M, Moilanen E, Suomalainen A, Lundbom N, Kaprio J, Rissanen A, Pietilainen KH. Characterising metabolically healthy obesity in weight-discordant monozygotic twins. Diabetologia. 2014 Jan;57(1):167-76. doi: 10.1007/s00125-013-3066-y. Epub 2013 Oct 8. PMID 24100782
- [Background] Jukarainen S, Heinonen S, Ramo JT, Rinnankoski-Tuikka R, Rappou E, Tummers M, Muniandy M, Hakkarainen A, Lundbom J, Lundbom N, Kaprio J, Rissanen A, Pirinen E, Pietilainen KH. Obesity Is Associated With Low NAD(+)/SIRT Pathway Expression in Adipose Tissue of BMI-Discordant Monozygotic Twins. J Clin Endocrinol Metab. 2016 Jan;101(1):275-83. doi: 10.1210/jc.2015-3095. Epub 2015 Nov 17. PMID 26574954
- [Background] Rappou E, Jukarainen S, Rinnankoski-Tuikka R, Kaye S, Heinonen S, Hakkarainen A, Lundbom J, Lundbom N, Saunavaara V, Rissanen A, Virtanen KA, Pirinen E, Pietilainen KH. Weight Loss Is Associated With Increased NAD(+)/SIRT1 Expression But Reduced PARP Activity in White Adipose Tissue. J Clin Endocrinol Metab. 2016 Mar;101(3):1263-73. doi: 10.1210/jc.2015-3054. Epub 2016 Jan 13. PMID 26760174
- [Background] Canto C, Houtkooper RH, Pirinen E, Youn DY, Oosterveer MH, Cen Y, Fernandez-Marcos PJ, Yamamoto H, Andreux PA, Cettour-Rose P, Gademann K, Rinsch C, Schoonjans K, Sauve AA, Auwerx J. The NAD(+) precursor nicotinamide riboside enhances oxidative metabolism and protects against high-fat diet-induced obesity. Cell Metab. 2012 Jun 6;15(6):838-47. doi: 10.1016/j.cmet.2012.04.022. PMID 22682224
- [Background] Trammell SA, Weidemann BJ, Chadda A, Yorek MS, Holmes A, Coppey LJ, Obrosov A, Kardon RH, Yorek MA, Brenner C. Nicotinamide Riboside Opposes Type 2 Diabetes and Neuropathy in Mice. Sci Rep. 2016 May 27;6:26933. doi: 10.1038/srep26933. PMID 27230286
- [Background] Airhart SE, Shireman LM, Risler LJ, Anderson GD, Nagana Gowda GA, Raftery D, Tian R, Shen DD, O'Brien KD. An open-label, non-randomized study of the pharmacokinetics of the nutritional supplement nicotinamide riboside (NR) and its effects on blood NAD+ levels in healthy volunteers. PLoS One. 2017 Dec 6;12(12):e0186459. doi: 10.1371/journal.pone.0186459. eCollection 2017. PMID 29211728